CLINICAL TRIAL: NCT06501092
Title: To Assess the Utility of the Point Mini in a Clinical Take-home Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Point Designs (Industry)
Collaborators: Children's Healthcare of Atlanta (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 445970; 4R44HD113485-02 (NIH)
Record Dates: First submitted 2024-07-05; First posted 2024-07-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Amputation; Traumatic, Hand; Amputation, Congenital
MeSH Terms: conditions — Amputation, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Current/No Device (No Intervention): Baseline outcome measurements will be performed with subject's existing partial hand prosthetic treatment, as deemed standard-of-care by the patient's prosthetist. Device types include, but are not limited to, no prosthesis, passive prosthesis, passive positional prosthesis, body-powered prosthesis, myoelectric prosthesis, or other assistive device.
- Point Mini (Experimental): Outcome measurements will be performed after the subject has been fit with a prosthesis at 3 different points in time: immediately post-fitting, ~30 days post-fitting, and ~60 days post-fitting.
  Interventions: Device: Point Mini

INTERVENTIONS:
Device: Point Mini — Patient is fit with the Point Mini finger prosthetic system, which consists of 1-4 ratcheting mechanical digits and mounting brackets
  Arms: Point Mini

SUMMARY:
The objective of this study is to evaluate the efficacy of the Point Mini system as compared to the subject's existing prosthetic treatment, which may include a prosthesis, other assistive device, or no device. This study will be a single subject crossover design where one group of 14 children with partial hand deficiencies will be evaluated on several metrics using their existing prosthetic treatment for one month and the Point Mini system for two months. Metrics include: in-clinic functional measures, subjective assessments, bilateral hand use, and prosthesis wear time.

ELIGIBILITY:
Inclusion Criteria:

* Partial hand loss with at least index and/or middle finger loss at the metacarpophalangeal (MCP) level
* Intact thumb with full range of motion
* Fluent in English
* Age between 5 and 15 years

Exclusion Criteria:

* Patients with a residual limb that is unhealed from the amputation surgery
* Unhealed wounds
* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon clinical evaluation
* Serious uncontrolled medical problems as judged by the project therapist

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ABILHAND-Kids | Baseline (pre-fitting)
  The ABILHAND-Kids is a measure of manual ability for children with upper limb impairment. ABILHAND-Kids consists of a questionnaire listing 21 manual activities and the child's parents respond with their perception of the child's performance and effort on a 3-point scale.
DISABKIDS | Baseline (pre-fitting)
  The DISABKIDS questionnaire measures general quality of life and the level of distress caused by the chronic condition. Both self-report and parent proxy-report versions are available. It is suitable for pediatric patients between 4-16 years of age with chronic health conditions.
ABILHAND-Kids | Immediately post-fitting
  The ABILHAND-Kids is a measure of manual ability for children with upper limb impairment. ABILHAND-Kids consists of a questionnaire listing 21 manual activities and the child's parents respond with their perception of the child's performance and effort on a 3-point scale.
DISABKIDS | Immediately post-fitting
  The DISABKIDS questionnaire measures general quality of life and the level of distress caused by the chronic condition. Both self-report and parent proxy-report versions are available. It is suitable for pediatric patients between 4-16 years of age with chronic health conditions.
ABILHAND-Kids | 30 days post-fitting
  The ABILHAND-Kids is a measure of manual ability for children with upper limb impairment. ABILHAND-Kids consists of a questionnaire listing 21 manual activities and the child's parents respond with their perception of the child's performance and effort on a 3-point scale.
DISABKIDS | 30 days post-fitting
  The DISABKIDS questionnaire measures general quality of life and the level of distress caused by the chronic condition. Both self-report and parent proxy-report versions are available. It is suitable for pediatric patients between 4-16 years of age with chronic health conditions.
ABILHAND-Kids | 60 days post-fitting
  The ABILHAND-Kids is a measure of manual ability for children with upper limb impairment. ABILHAND-Kids consists of a questionnaire listing 21 manual activities and the child's parents respond with their perception of the child's performance and effort on a 3-point scale.
DISABKIDS | 60 days post-fitting
  The DISABKIDS questionnaire measures general quality of life and the level of distress caused by the chronic condition. Both self-report and parent proxy-report versions are available. It is suitable for pediatric patients between 4-16 years of age with chronic health conditions.

SECONDARY OUTCOMES:
Weekly Diary Entries | Through study completion, an average of 3 months
  Throughout the study, subjects and their parents will fill out weekly logs asking their experiences during the day, number of hours wearing the device, descriptions of the tasks performed, and open-response sections to clarify/detail any other events. The weekly logs will be in sealed envelopes and not opened until the completion of the study by the experimenters.

CONTACTS AND LOCATIONS:
Overall Officials: Levin Sliker, PhD, Principal Investigator — Point Designs
Locations (2):
- United States (2):
  - Point Designs, Lafayette, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No